CLINICAL TRIAL: NCT02262403
Title: Study of Immuno-regulatory Mechanisms Induced by Hookworm Infection
Brief Title: Hookworm Immune Regulation Project
Acronym: HIRP-01
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Brugmann University Hospital (Other)
Collaborators: Université Libre de Bruxelles (Other)
Responsible Party: Principal Investigator, Olivier Michel, Head of clinic, Brugmann University Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CHUB-HIRP-01
Record Dates: First submitted 2014-09-16; First posted 2014-10-13 (Estimated); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Hookworm Infection
Keywords: Hookworm; Helminths; Treg; Immune regulation; Vietnam; Allergic diseases
MeSH Terms: conditions — Hookworm Infections; Ancylostomiasis | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hookworm infected (Experimental): The amount, phenotype and function of Treg will be explored at several time points. Cultures with environmental antigen will be subsequently performed.
  Interventions: Other: Blood and feces sampling
- Non infected (hookworms) healthy subjects (Active Comparator): All the tests done in the experimental hookworm infected group will be also done in the comparator non infected group.
  Interventions: Other: Blood and feces sampling

INTERVENTIONS:
Other: Blood and feces sampling — Blood and feces samples will be examined after 14 days, 28 days, 3 months and 16 months. This will require blood and feces sampling. The study is therefore defined as 'interventional' rather than 'observational' as it includes acts outside the standard of care.

SUMMARY:
The main objective of this study is to characterize the regulatory immune response induced by hookworm in an infected Vietnamese rural population from the periphery of HCM, evolution after infection treatment and during potential naturally reinfection.

DETAILED DESCRIPTION:
Population: 20 healthy adults (18-65 years) infected and non infected by Hookworm will be recruited and treated according to Good Clinical Practice recommendations.

Allergy will be excluded by skin prick tests. Amount and phenotype of Treg will be explored at several time points. Subsequent culture with environmental antigen will be performed on cryopreserved cells.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old adults in good health status
* To live in rural regions at risk of soil transmitted helminthes
* Hookworm infection (infected group)
* Uninfected by Hookworms (control group)

Exclusion Criteria:

* Pregnant woman
* Positive allergic history
* Auto-immune and/or HIV disease
* Antihelminthics drug in the last 6 months and other current parasitic infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2014-08-01 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Amount and phenotype of Treg | 0-12 weeks
  Four colors flow cytometry Treg measurements and phenotyping (FACSCantoII).

OTHER OUTCOMES:
PBMC culture and cryopreservation | after 12 weeks
  Assessment of the orientation of the adaptative immune response to Dermatophagoides pteronyssinus.Subsequent Treg function testing and cell cultures (with environmental antigen) on cryopreserved PBMC (Peripheral Blood Mononuclear cells).

CONTACTS AND LOCATIONS:
Overall Officials: Virginie Doyen, MD, Principal Investigator — CHU Brugmann - ULB
Locations (1):
- Pham Ngoc Thach University of Medecine, Ho Chi Minh City, Distict 10, Vietnam

REFERENCES:
- [Background] Flohr C, Tuyen LN, Quinnell RJ, Lewis S, Minh TT, Campbell J, Simmons C, Telford G, Brown A, Hien TT, Farrar J, Williams H, Pritchard DI, Britton J. Reduced helminth burden increases allergen skin sensitization but not clinical allergy: a randomized, double-blind, placebo-controlled trial in Vietnam. Clin Exp Allergy. 2010 Jan;40(1):131-42. doi: 10.1111/j.1365-2222.2009.03346.x. Epub 2009 Sep 15. PMID 19758373
- [Background] Flohr C, Tuyen LN, Lewis S, Quinnell R, Minh TT, Liem HT, Campbell J, Pritchard D, Hien TT, Farrar J, Williams H, Britton J. Poor sanitation and helminth infection protect against skin sensitization in Vietnamese children: A cross-sectional study. J Allergy Clin Immunol. 2006 Dec;118(6):1305-11. doi: 10.1016/j.jaci.2006.08.035. Epub 2006 Oct 13. PMID 17157661
- [Background] Finlay CM, Walsh KP, Mills KH. Induction of regulatory cells by helminth parasites: exploitation for the treatment of inflammatory diseases. Immunol Rev. 2014 May;259(1):206-30. doi: 10.1111/imr.12164. PMID 24712468
- [Background] Sakaguchi S, Vignali DA, Rudensky AY, Niec RE, Waldmann H. The plasticity and stability of regulatory T cells. Nat Rev Immunol. 2013 Jun;13(6):461-7. doi: 10.1038/nri3464. Epub 2013 May 17. PMID 23681097